CLINICAL TRIAL: NCT03246347
Title: A Phase II Trial of Androgen Deprivation, Docetaxel and Enzalutamide in Patients With Metastatic Hormone Sensitive Prostate Cancer
Brief Title: A Trial of Androgen Deprivation, Docetaxel, and Enzalutamide for Metastatic Prostate Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Astellas Pharma Inc (Industry); Medivation, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00081385; LCI-GU-PRO-ADDE-001 (Other: Atrium Health); Pro00018087 (Other: Wake Forest University Health Sciences)
Record Dates: First submitted 2017-08-04; First posted 2017-08-11 (Actual); Results first posted 2023-09-22 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Prostate Cancer; Prostate Adenocarcinoma
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Docetaxel; enzalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single Arm (Experimental): Docetaxel + Enzalutamide + Androgen Deprivation Therapy
  Interventions: Drug: ADT+Docetaxel+Enzalutamide

INTERVENTIONS:
Drug: ADT+Docetaxel+Enzalutamide — combination therapy as listed above
  Other Names: Taxotere; Xtandi

SUMMARY:
This is a study with the combination of androgen deprivation therapy (ADT) and docetaxel with the addition of enzalutamide in the treatment of subjects with metastatic prostate cancer. The purpose of this study is to assess if ADT + docetaxel + enzalutamide is well tolerated and demonstrates improved efficacy compared to ADT + docetaxel.

DETAILED DESCRIPTION:
This is a single center, single arm, phase II trial designed to evaluate the 12 month PSA complete response rate in patients with metastatic hormone sensitive prostate cancer treated with ADT, docetaxel and enzalutamide. The primary endpoint of this study will be 12-month PSA complete response rate, which will be assessed against a contemporary historical control rate for the combination of ADT and docetaxel alone in the metastatic hormone naive setting. The study will be conducted at all participating sites across North and South Carolina within the Levine Cancer Institute network. Enrollment is anticipated to be completed within 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the prostate without evidence of small cell carcinoma or greater than 50% neuroendocrine differentiation. Metastatic disease must be present including soft tissue, and/or bone metastases OR nonregional lymph node involvement prior to study enrollment. If the subject has regional lymph node involvement, there must be at least one additional site of disease including visceral, non-regional nodal or skeletal metastases.
* ADT with surgical castration with bilateral orchiectomy or medical castration with LHRH agonist or LHRH antagonist therapy may have been initiated no greater than 112 days (16 weeks) prior to enrollment date. Subjects who initiated ADT prior to consent, are not eligible if PSA has risen ≥ 25% and ≥ 2 ng/ml above nadir value since initiation of ADT prior to consent.
* At least one PSA level of ≥ 5 ng/ml within 90 days prior to consent.
* Prior ADT for non-metastatic disease with LHRH agonist or LHRH antagonist therapy in the neoadjuvant/adjuvant setting is permitted if:

  1. Total duration of therapy did not exceed 36 months
  2. 6 months have elapsed since completion of therapy prior to consent,
  3. Serum testosterone > 50 ng/dl within 28 days prior to reinitiation of ADT for metastatic disease
  4. Prior ADT for non-metastatic disease must have accompanied definitive local therapy for curative intent.
* Age ≥ 18 years.
* ECOG performance status 0-2.
* Adequate liver function: AST and ALT <1.5x upper limit of normal, total bilirubin < 1x upper limit of normal.
* Adequate bone marrow function: Platelets >100,000 cells/mm3, Hemoglobin > 8.0g/dL and ANC > 1,500 cells/mm3.
* Adequate renal function with a creatinine clearance (based on Cockcroft-Gault formula) ≥ 30 mL/min.
* Ability to understand and the willingness to sign a written informed consent document.
* Able to swallow and retain oral medication

Exclusion Criteria:

* Personal history of seizure.
* Personal history of conditions that may predispose to seizure activity including cortical cerebrovascular accident or brain trauma.
* Known central nervous system metastases, including involvement of brain parenchyma and leptomeninges.
* Personal history of any condition that may impair absorption of enzalutamide.
* Prior or current therapy with ketoconazole, abiraterone, enzalutamide, apalutamide (ARN-509, JNJ-56021927), darolutamide (ODM-201, BAY1841788) or cytotoxic chemotherapy such as docetaxel, cabazitaxel, cyclophosphamide.
* Prior therapy with bicalutamide, nilutamide or flutamide within 14 days of enrollment.
* Within 28 days of major surgery and/or lack of recovery from prior surgical procedure or 14 days of palliative radiation prior to enrollment.
* Prior or current therapy with an investigational agent for metastatic prostate cancer.
* Known hypersensitivity to drugs formulated with polysorbate 80.
* Personal history of posterior reversible encephalopathy syndrome.
* CTCAE version 4.0 grade 2-4 peripheral sensory neuropathy.
* Human immunodeficiency virus infection or active hepatitis B or C infection.
* Uncontrolled and current illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements in the opinion of the investigator.
* Presence of any of the following within the previous 3 months prior to enrollment: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, congestive heart failure, or cerebrovascular accident including transient ischemic attack.
* History of an additional active malignancy within 12 months prior to the date of consent (except non-melanoma skin cancer).
* Current use of strong CYP2C8 inhibitors, CYP3A4 inducers or CYP3A4, CYP2C9 or CYP2C19 substrates with a narrow therapeutic range as listed in Section 7.2.1.
* Any condition that requires the use of prednisone > 10mg daily, or equivalent daily glucocorticoid dose, for greater than 14 days

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-08-23 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2028-03 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Earle Burgess, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Levine Cancer Institute, Charlotte, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Single Arm
Started | 40
Completed | 17 (At the time of reporting for the primary objective, seventeen subjects have completed the study. Reasons for completion include death (N=13), consent withdrawal (N=3), and loss to follow-up (N=1). Twenty-three subjects remain on study and data is still captured.)
Not Completed | 23
Not completed — On Study | 23

BASELINE CHARACTERISTICS:
Population: All enrolled patients (i.e., patients initiating enzalutamide and docetaxel)
Arm/Group | Single Arm
Number analyzed (Participants) | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 25
  >=65 years | 15
Age, Continuous [Mean (Full Range); unit: years] | 64.95 [51 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 40
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 14
  White | 26
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 40
Disease volume at enrollment [Count of Participants; unit: Participants]
  Low volume | 10
  High volume | 30

OUTCOME MEASURES:

1. Primary Outcome: 52-week PSA Complete Response (CR) Rate
Description: The 52-week PSA CR rate was defined as the proportion of participants achieving PSA complete response (CR) at 52-weeks (+/- 1 week) from date of enrollment (i.e., initiation of both enzalutamide and docetaxel) of all evaluable participants. PSA CR was defined as PSA level less than 0.2 ng/ml for two consecutive measurements at least three weeks apart (date of initial PSA level 0.2 ng/ml was acknowledged as date of response). In subjects with missed PSA assessments at 52 (+/- 1) weeks, (a) if a confirmed CR was achieved and at least one PSA assessment occurred beyond the 52-week window showed serologic complete response (providing the subject did not earlier experience confirmed progressive disease), the subject achieved 52-week PSA Complete Response and (b) if confirmed CR was achieved before the 52-week window and the first assessment after the 52-week window was not a CR, the subject did not achieve a 52-week PSA Complete Response.
Time Frame: 52 weeks
Population: The evaluable population for the primary analysis included subjects who began study treatment and did not discontinue enzalutamide prior to the development of castrate resistance for reasons other than can be attributed to study treatment. Four enrolled subjects were not evaluable for the analysis of the primary objective for reasons including consent withdrawal and noncompliance.
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 36
Participants | 22
Statistical Analysis 1: Comparison: Single Arm; The 12-month PSA CR rate with ADT + docetaxel is 27.7% (Sweeney 2015); we estimated that the lower limit of the 95% CI was 23.4%. We sought to test the null hypothesis that the 52-week PSA CR rate for subjects treated with study therapy was <=25%. We anticipated enrolling 39 subjects and this design would provide 90% power with a 1-sided alpha =0.10 significance level, assuming the true 52-week PSA CR rate was 45%. An improvement from 25% to 45% in 52-week PSA CR rate was considered important; Test type: Superiority; p < 0.001, One-sided test for binomial proportions; Proportion = .6111, 95% CI 2-sided [.4346 to .7686]

2. Secondary Outcome: Serologic Response Rate
Time Frame: Duration of study participation, an average of 2 years
Reporting Status: Not Posted

3. Secondary Outcome: Radiographic Response Rate
Time Frame: Duration of study participation, an average of 2-3 years
Reporting Status: Not Posted

4. Secondary Outcome: Time to Castrate Resistance
Time Frame: Duration of study participation, an average of 2 years
Reporting Status: Not Posted

5. Secondary Outcome: Serologic Progression Free Survival
Time Frame: Duration of study participation, an average of 2 years
Reporting Status: Not Posted

6. Secondary Outcome: Radiographic Progression Free Survival
Time Frame: Duration of study participation, an average of 2-3 years
Reporting Status: Not Posted

7. Secondary Outcome: Overall Survival
Time Frame: Duration of study participation, an average of 5 years
Reporting Status: Not Posted

8. Secondary Outcome: Time to Treatment Failure
Time Frame: Duration of study participation, an average of 2-3 years
Reporting Status: Not Posted

9. Secondary Outcome: Treatment-related Adverse Events as Assessed by CTCAE v4.0
Time Frame: Duration of study participation, an average of 5 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events are collected from initiation of study drugs to 30 days following cessation of study drugs. The maximum adverse event collection timeframe was 5.8 years.
Description: Treatment-emergent adverse events were reported and defined as an adverse event that occurred after treatment start that was not present at the time of treatment start or an adverse event that increased in severity after treatment start if the event was present at the time of treatment start.
Arm/Group | Single Arm
All-Cause Mortality (participants affected / at risk) | 13/40
Serious Adverse Events (participants affected / at risk) | 14/40
Other Adverse Events (participants affected / at risk) | 40/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm (N=40)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 1 (1)
ATRIAL FLUTTER (Cardiac disorders) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
CARDIAC DISORDERS - OTHER, ICD Read Malfunction (Cardiac disorders) | 1 (1)
COLITIS (Gastrointestinal disorders) | 1 (2)
CONFUSION (Psychiatric disorders) | 1 (1)
DEHYDRATION (Metabolism and nutrition disorders) | 1 (2)
DYSPHAGIA (Gastrointestinal disorders) | 1 (1)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 1 (1)
ENCEPHALOPATHY (Nervous system disorders) | 2 (2)
ESOPHAGEAL INFECTION (Infections and infestations) | 1 (1)
FALL (Injury, poisoning and procedural complications) | 2 (2)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 2 (2)
FEVER (General disorders) | 1 (1)
GASTROINTESTINAL DISORDERS - OTHER, Pneumoperitoneum (Gastrointestinal disorders) | 2 (2)
GENERALIZED MUSCLE WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 (1)
HIP FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPOGLYCEMIA (Metabolism and nutrition disorders) | 1 (1)
INFECTIONS AND INFESTATIONS - OTHER, Bacteremia (Infections and infestations) | 1 (1)
INJURY, POISONING AND PROCEDURE COMPLICATIONS - OTHER, MVA (Injury, poisoning and procedural complications) | 1 (1)
KIDNEY INFECTION (Infections and infestations) | 1 (1)
LUNG INFECTION (Infections and infestations) | 1 (1)
MULTI-ORGAN FAILURE (General disorders) | 1 (2)
MUSCLE WEAKNESS RIGHT-SIDED (Musculoskeletal and connective tissue disorders) | 1 (1)
NEOPLASMS BENIGN, MALIGNANT AND UNSPECIFIED - OTHER, Urothelial Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
NEUTROPHILL COUNT DECREASED (Investigations) | 1 (1)
NON-CARDIAC CHEST PAIN (General disorders) | 1 (1)
SEPSIS (Infections and infestations) | 1 (1)
STROKE (Nervous system disorders) | 1 (1)
URETHRAL INFECTION (Infections and infestations) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1)
URINARY TRACT OBSTRUCTION (Renal and urinary disorders) | 1 (2)
WHITE BLOOD CELL DECREASED (Investigations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Single Arm (N=40)
ABDOMINAL PAIN (Gastrointestinal disorders) | 6
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 4
ALKALINE PHOSPHATASE INCREASED (Investigations) | 4
ALLERGIC RHINITIS (Respiratory, thoracic and mediastinal disorders) | 5
ALOPECIA (Skin and subcutaneous tissue disorders) | 16
ANEMIA (Blood and lymphatic system disorders) | 4
ANOREXIA (Metabolism and nutrition disorders) | 9
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 13
BACK PAIN (Musculoskeletal and connective tissue disorders) | 5
BONE PAIN (Musculoskeletal and connective tissue disorders) | 4
CONSTIPATION (Gastrointestinal disorders) | 4
COUGH (Respiratory, thoracic and mediastinal disorders) | 9
DEPRESSION (Psychiatric disorders) | 3
DIARRHEA (Gastrointestinal disorders) | 13
DIZZINESS (Nervous system disorders) | 8
DRY EYE (Eye disorders) | 3
DRY SKIN (Skin and subcutaneous tissue disorders) | 3
DYSGEUSIA (Nervous system disorders) | 16
DYSPHAGIA (Gastrointestinal disorders) | 3
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 10
EDEMA LIMBS (General disorders) | 12
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 3
FALL (Injury, poisoning and procedural complications) | 5
FATIGUE (General disorders) | 32
FLU LIKE SYMPTOMS (General disorders) | 3
GASTROESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 3
GENERALIZED MUSCLE WEAKNESS (Musculoskeletal and connective tissue disorders) | 8
GYNECOMASTIA (Reproductive system and breast disorders) | 4
HEADACHE (Nervous system disorders) | 7
HEMATURIA (Renal and urinary disorders) | 4
HOT FLASHES (Vascular disorders) | 13
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 4
HYPERTENSION (Vascular disorders) | 5
HYPOKALEMIA (Metabolism and nutrition disorders) | 3
HYPOTENSION (Vascular disorders) | 5
INFECTIONS AND INFESTATIONS - OTHER, SPECIFY: COVID-19 (Infections and infestations) | 8
INFUSION RELATED REACTION (General disorders) | 3
INSOMNIA (Psychiatric disorders) | 9
LUNG INFECTION (Infections and infestations) | 4
MUCOSITIS ORAL (Gastrointestinal disorders) | 3
MUSCLE WEAKNESS LOWER LIMB (Musculoskeletal and connective tissue disorders) | 3
MYALGIA (Musculoskeletal and connective tissue disorders) | 4
NAIL DISCOLORATION (Skin and subcutaneous tissue disorders) | 11
NAIL INFECTION (Infections and infestations) | 3
NAIL LOSS (Skin and subcutaneous tissue disorders) | 6
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 4
NAUSEA (Gastrointestinal disorders) | 14
NERVOUS SYSTEM DISORDERS - OTHER, SPECIFY: RESTLESS LEG SYNDROME (Nervous system disorders) | 3
NEUTROPHIL COUNT DECREASED (Investigations) | 6
NON-CARDIAC CHEST PAIN (General disorders) | 4
ORAL PAIN (Gastrointestinal disorders) | 3
PAIN (General disorders) | 10
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 8
PARESTHESIA (Nervous system disorders) | 5
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 18
SORE THROAT (Respiratory, thoracic and mediastinal disorders) | 3
TOOTHACHE (Gastrointestinal disorders) | 3
UPPER RESPIRATORY INFECTION (Infections and infestations) | 5
URINARY FREQUENCY (Renal and urinary disorders) | 6
URINARY RETENTION (Renal and urinary disorders) | 3
URINARY TRACT INFECTION (Infections and infestations) | 4
VERTIGO (Ear and labyrinth disorders) | 3
VOMITING (Gastrointestinal disorders) | 8
WATERING EYES (Eye disorders) | 6
WEIGHT GAIN (Investigations) | 8
WEIGHT LOSS (Investigations) | 5
WHITE BLOOD CELL DECREASED (Investigations) | 4
DYSPEPSIA (Gastrointestinal disorders) | 3
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-03-14): https://cdn.clinicaltrials.gov/large-docs/47/NCT03246347/Prot_SAP_001.pdf
  • Informed Consent Form (2022-06-06): https://cdn.clinicaltrials.gov/large-docs/47/NCT03246347/ICF_000.pdf